CLINICAL TRIAL: NCT02383953
Title: Non Genetic Factors in the Pathogenesis of Inflammatory Bowel Disease in Twins
Brief Title: SSAT 054: Non Genetic Factors in the Pathogenesis of IBD in Twins
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SSAT 054
Record Dates: First submitted 2015-01-07; First posted 2015-03-10 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: twins; IBD; UC; CD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (plasma), stool, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate the role of non-genetic factors in the pathogenesis of inflammatory bowel disease.An exploratory study to investigate differences between the epigenome, microbiota and functional immunology in twins discordant for inflammatory bowel disease.

DETAILED DESCRIPTION:
Background: The inflammatory bowel diseases (IBD), Crohn's Disease (CD) and Ulcerative Colitis (UC), are debilitating conditions with a complex aetiology. The biggest risk factor for developing IBD is having an affected first degree relative. However when an identical twin is diagnosed with IBD, the other twin goes on to develop the condition in only 20-55% of cases.

Recent research suggests the microbiota the ecosystem of bacteria within the gut may trigger disease in susceptible individuals. Another important research area is the epigenome changes to the structure and regulation of our genome which occur throughout our life. It is known that siblings of Crohn's Disease sufferers have a changes to the immune system characteristic of Crohn';s. However it is not known whether these changes are due to genetic similarity or shared environment. Comparison between mono and dizygotic twins elucidates the relative importance of genetic and environmental factors.

Primary Objective: An exploratory study to investigate differences between the epigenome, microbiota and functional immunology in twins discordant for inflammatory bowel disease.

Study Design: Multicentre basic science study involving human participants

Planned sample size: 200 data subjects (100 twin pairs)

Methodology:

A) Identification of twin pairs where one or both have inflammatory bowel disease via:

1. IBD Nixon Twin and Multiplex Registry.
2. Advertising for twin pairs via BSG website and newsletters/patient support groups/social media sites/clinic posters.
3. Identification by study sites B) Obtaining formal written consent C) Collection of blood, stool and urine.

D) The following analysis will be carried out:

* Epigenetics (blood) DNA extraction and subsequent methylation analysis and bisulphate conversion with 450 Illumina beadchip assay
* Functional immunology (blood) - flow cytometry of CD3, CD4 and CD8 cells. (London Twin pairs discordant for Crohn's Disease)
* 16S rRNA gene sequencing (stool) - of bacterial DNA
* Metabolomic profiling (Urine and stool) - using Nuclear Magnetic Resonance (NMR) and mass spectrometry E) Collection of dietary history information for the previous 72hr period Study Duration: 2 years (single visit).

ELIGIBILITY:
Inclusion Criteria:

* Monozygotic twins discordant for IBD
* Monozygotic twins concordant for IBD
* Dizygotic twins discordant for IBD
* Dizygotic twins concordant for IBD
* Healthy controls

Exclusion Criteria:

* <18 years old
* Antibiotics within past 3 months of sample collection
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Difference in DNA methylation patterns between twin pairs | 1 day (1 visit only)
Difference in microbiota composition and metabolomic profiles between IBD phenotypes | 1 day (1 visit only)
Comparison of microbiota composition and metabolic profiles with DNA methylation patterns | 1 day (1 visit only)
Difference in T cell phenotypes and antigen presenting cells between twin pairs discordant for IBD | 1 day (1 visit only)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Harbord, MD, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- Chelsea and Westminster Hosptial, London, United Kingdom